CLINICAL TRIAL: NCT00758368
Title: Comparison of Continuous and Pulsatile Apomorphine Administration in Parkinson's Disease Complicated by Levodopa-induced Dyskinesia
Brief Title: Comparison of Continuous and Pulsatile Apomorphine in Parkinson's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate support to conduct the study
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John G. Nutt, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS021062-21 (NIH); R01NS021062-21 (NIH); eIRB 2167 (Other: Oregon Health and Science University)
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; PD; pulsatile apomorphine; dyskinesia; apomorphine; continuous dopaminergic stimulation
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulatory Pump (Experimental): Participants will receive apomorphine via a pump. Participants in the Continuous Delivery Arm will self-administer apomorphine continuously (12-14 hours a day) using a portable pump.
  Interventions: Drug: Apomorphine
- Subcutaneous Injections (Active Comparator): Participants will receive apomorphine via an injection pen. Participants in the Intermittent Delivery Arm will self-administer apomorphine at intervals, via a injection, using pen injector.
  Interventions: Drug: Apomorphine

INTERVENTIONS:
Drug: Apomorphine — Participants in both arms will receive the study drug apomorphine for 6 months. One group will receive it continuously using a portable pump during waking hours, and the other group will receive it intermittently by bolus injections. The continuous delivery group will receive up to 100 mg apomorphine per 24 hours, delivered subcutaneously by ambulatory pump. The intermittent delivery group will receive up to 5 subcutaneous injections totaling up to 20 mg daily.
  Other Names: Apokyn, apomorphine, apo-go pump

SUMMARY:
The purpose of this study is to compare the effects of apomorphine, given by two different methods, to determine how best to manage dyskinesias.

DETAILED DESCRIPTION:
Levodopa is a drug that can be taken by mouth, and improves the symptoms of Parkinson's disease (PD). However it can eventually cause involuntary movements called dyskinesia and motor fluctuations-fluctuations in the control of symptoms, often referred to as "off" and "on." Apomorphine is a drug that works as well as levodopa, but does not work if taken by mouth.

The purpose of this study is to compare the effects of apomorphine in people with PD who have levodopa-induced motor fluctuations and dyskinesias. In the trial, researchers will compare the effects of apomorphine administered by subcutaneous bolus injections (pulsatile) and by ambulatory infusion pumps (continuous) in 24 people with PD, for 6 months.

After an initial screening, potential participants will undergo a test to verify that they can tolerate and respond to apomorphine. Those who meet all of the requirements will be randomized to receive the study drug via injections (shots) using an injector pen or a portable infusion pump. Apomorphine will be given either continuously using the portable pump during the waking day or intermittently by injection, for 6 months. The pump will be carried on a belt and connected by a tube to a small needle under the skin. Injections of apomorphine under the skin will be self-administered by the participants or administered by friends or family members using injector pens.

After 6 months, the effects of apomorphine use will be assessed by measuring how the participants respond to levodopa and by measuring their symptoms during the course of the study. Participants will be followed initially every week, then biweekly, and then monthly in an outpatient clinic for 6 months. During this time, they may receive adjustments of apomorphine doses as well as doses of other antiparkinson medications.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's Disease
* clear response to levodopa (sinemet)
* "off" at least 20% of waking day
* dyskinesias present for at least two hours of waking day
* subject or caregiver able to master use of drug delivery system (injector pen or pump)

Exclusion Criteria:

* physical complications that would preclude safe participation
* standing systolic BP of <80
* lack of tolerance or response to apomorphine
* drug/alcohol abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in dyskinesia severity and duration during the levodopa infusion, measured with a clinical rating scale during two-hour levodopa infusion | at baseline and after 6 months

SECONDARY OUTCOMES:
Improvement in motor performance, measured as change in tapping speed during levodopa infusion | at baseline and after 6 months
Improvement in "on" time, as measured by subject diaries | at baseline and after 6 months
Reduction in levodopa and adjunct drug use | at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John G. Nutt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Manson AJ, Turner K, Lees AJ. Apomorphine monotherapy in the treatment of refractory motor complications of Parkinson's disease: long-term follow-up study of 64 patients. Mov Disord. 2002 Nov;17(6):1235-41. doi: 10.1002/mds.10281. PMID 12465062
- [Background] Stocchi F, Ruggieri S, Vacca L, Olanow CW. Prospective randomized trial of lisuride infusion versus oral levodopa in patients with Parkinson's disease. Brain. 2002 Sep;125(Pt 9):2058-66. doi: 10.1093/brain/awf214. PMID 12183351
- [Background] Stocchi F, Vacca L, Ruggieri S, Olanow CW. Intermittent vs continuous levodopa administration in patients with advanced Parkinson disease: a clinical and pharmacokinetic study. Arch Neurol. 2005 Jun;62(6):905-10. doi: 10.1001/archneur.62.6.905. PMID 15956161